CLINICAL TRIAL: NCT03072940
Title: 3 T Multimodal MRI in Idiopathic RBD
Brief Title: Brain Imaging in the Idiopathic REM Sleep Behavior Disorder (ALICE)
Acronym: ALICE
Status: Completed | Type: Observational
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Collaborators: NRJ Foundation - Institute of France (Unknown); National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: ADOREPS_7
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: REM Sleep Behavior Disorder; Healthy
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with idiopathic RBD
  Interventions: Other: Clinical investigations
- Healthy volunteers
  Interventions: Other: Clinical investigations

INTERVENTIONS:
Other: Clinical investigations — Clinical examination, motor, cognitive, autonomous, psychological, olfactory and color vision tests, and rapid eye movement sleep characterization using video-polysomnography and 3 T magnetic resonance imaging

SUMMARY:
Idiopathic rapid eye movement sleep behavior disorder (iRBD) is characterized by nocturnal violence, increased muscle tone during REM sleep and the lack of any other neurological disease. However, iRBD can precede parkinsonism and dementia by several years. The causes of the loss of muscle atonia during REM sleep in these patients are unclear. Using 3 T MRI and neuromelanin- sensitive sequences, the signal intensity was previously found to be reduce in the locus coeruleus/subcoeruleus area of patients with Parkinson's disease and RBD. Here, the investigators aimed at studying the integrity of the locus coeruleus/ subcoeruleus complex with neuromelanin-sensitive imaging in 21 patients with iRBD and compared the results with those from 21 age- and gender-matched healthy volunteers. All subjects will undergo a clinical examination, motor, cognitive, autonomous, psychological, olfactory and color vision tests, and rapid eye movement sleep characterization using video-polysomnography and 3 T magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

- idiopathic RBD (criteria of the international classification of sleep disorders-3)

For healthy controls : no neurologic or psychiatric disorder

Exclusion Criteria:

* Contraindication to MRI
* Do not speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Signal in the subcoeruleus/coeruleus complex | 24h
  Brain imaging signal in the subcoeruleus/coeruleus complex in 3T multimodal MRI, using neuromelanin-sensitive sequence

SECONDARY OUTCOMES:
Substantia nigra quantity | 24h
  size of the substantia nigra
Quality of Sleep | 24h
  Measures in videopolysomnography of efficiency of sleep
Cognition | 24h
  Cognition status (MoCA test)
Olfactory function | 24h
  Olfactory function (sniff test)
Color vision | 24h
  Color vision function

CONTACTS AND LOCATIONS:
Locations (1):
- Pitie Salpetriere hospital, Paris, France

REFERENCES:
- [Result] Ehrminger M, Latimier A, Pyatigorskaya N, Garcia-Lorenzo D, Leu-Semenescu S, Vidailhet M, Lehericy S, Arnulf I. The coeruleus/subcoeruleus complex in idiopathic rapid eye movement sleep behaviour disorder. Brain. 2016 Apr;139(Pt 4):1180-8. doi: 10.1093/brain/aww006. Epub 2016 Feb 26. PMID 26920675